CLINICAL TRIAL: NCT02216565
Title: Benefits of the Endovascular Treatment in the Early Management of Proximal Sylvian Artery Thrombosis in Patients Refractory or Ineligible to Intravenous Fibrinolysis : a Multicenter Controled Randomized Trial
Brief Title: Embolectomy in Acute SYlvian Thrombosis in Refractory or Ineligible Patients to ALteplase
Acronym: EASY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After results of other studies published : EASY study became lapsed
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A00519-38
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Stroke, Acute
Keywords: Stroke; Endovascular treatment; Tandem carotid occlusions; Fibrinolysis
MeSH Terms: conditions — Stroke | interventions — Hospitalization; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical treatment (Other): Conventional medical non-interventional treatment
  Interventions: Other: Hospitalization in specialized neuro-vascular unit; Drug: Alteplase if patient is eligible; Other: Supportive care
- Endovascular treatment (Other): Conventional medical treatment plus endovascular treatment
  Interventions: Other: Hospitalization in specialized neuro-vascular unit; Drug: Alteplase if patient is eligible; Other: Supportive care; Procedure: Endovascular treatment

INTERVENTIONS:
Other: Hospitalization in specialized neuro-vascular unit
Drug: Alteplase if patient is eligible — Alteplase intravenous thrombolysis performed if patient is eligible (if not contraindicated)
Other: Supportive care — Drugs, procedures and techniques aimed at preventing/managing complications or aggravation of the patient's neurological condition
Procedure: Endovascular treatment — Recanalization treatment (thrombectomy / intraarterial thrombolysis)
  Arms: Endovascular treatment

SUMMARY:
This trial aims at comparing two strategies currently used to address acute ischemic stroke of the middle cerebral artery : medical treatment without endovascular treatment on the one hand, and medical treatment plus endovascular treatment on the other hand. The efficiency of the strategies will be assessed in terms of early neurological clinical recovery.

The study will focus on three particular situations : (1) tandem internal carotid and middle cerebral artery occlusion, (2) situations where patient cannot benefit from fibrinolysis because of high risk of haemorrhage, (3) situations where fibrinolysis is not recommended because of a delay superior to 4.5 hours.

The hypothesis to be tested is that medical approach plus endovascular treatment is superior to medical treatment alone

ELIGIBILITY:
Inclusion Criteria:

* Radiologically proven acute proximal occlusion of middle cerebral artery

AND one of the three following :

1. tandem internal carotid / middle cerebral artery occlusion
2. intravenous thrombolysis contraindicated because of high risk of haemorrhage
3. intravenous thrombolysis not possible because of delay > 4.5 hours

Exclusion Criteria:

* Impossibility to perform endovascular recanalization within 6h
* Clinically minor stroke (NIHSS score below 5 at baseline)
* Extended cerebral infarction
* Severe comorbidity
* Life expectancy below 3 months before stroke
* Pregnancy or breastfeeding
* modified Rankin Score superior to 2 before stroke

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-08-31 (Actual); Study Completion 2017-08-24 (Actual)

PRIMARY OUTCOMES:
Improvement in NIHSS score after 24h | 24 hours
  Percentage of improvement in the National Institute of Health Stroke Score (NIHSS) between baseline (t0) and h24 (t1) calculated as follow :
  [NIHSS(t0) - NIHSS(t1)] / NIHSS(t0)

SECONDARY OUTCOMES:
Improvement in NIHSS score after 7 days | 7 days
  Percentage of improvement in the National Institute of Health Stroke Score (NIHSS) between baseline (t0) and day7 (t2) calculated as follow :
  [NIHSS(t0) - NIHSS(t2)] / NIHSS(t0)
Functional recovery after 3 months | 3 months
  modified Rankin Score (mRS) after 3 months ("positive recovery" if mRS <=2, "excellent recovery" if mRS<=1)
Fatality within 7 days | 7 days
  Proportion of patients deceased within seven days after stroke
Fatality within 3 months | 3 months
  Proportion of patients deceased within 3 months after stroke

CONTACTS AND LOCATIONS:
Overall Officials: Marc-Antoine Labeyrie, MD, Principal Investigator — Hopital Lariboisiere, Paris; Michel Piotin, MD, Principal Investigator — Fondation Ophtalmologique Adolphe de Rothschild, Paris
Locations (3):
- France (3):
  - Hopital Henri Mondor, Créteil
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hopital Foch, Suresnes